Official title: Examining the Association of Sun Salutations and Aerobic Exercise With Cognition Among Adults With Psychosocial Stress

NCT number: NCT04077645

Document date: November 8, 2021

Data were analyzed in SPSS v.27. Data were checked for outliers (±2.5 standard deviations from the mean) and winzorized, i.e., values + - 2.5 standard deviations from the mean were replaced with the highest or lowest present value in the dataset. Five outliers in TMT and one outlier in reaction time for 2-back non-match task were winzorized. There was no missing data. A 2 (time) x 3 (group) repeated measures analysis of covariance (ANCOVA) was conducted for n-back, TMT, and DSST. Covariates included baseline score, pulse pressure, estimated cardiorespiratory fitness, and education. A univariate ANCOVA was conducted for psychosocial measures, accounting for baseline scores. Bonferroni adjustment was used for post-hoc comparisons, and the alpha level was set at .05. Partial eta squared (ηp2) was used as the effect size (.05 or smaller = small, .06 = medium, .14 = large) (Olejnik & Algina, 2000).